CLINICAL TRIAL: NCT03386864
Title: Metabolic Determinants of Cardiac Function
Status: Completed | Type: Observational
Sponsor: German Diabetes Center (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 5263R
Record Dates: First submitted 2017-05-29; First posted 2017-12-29 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure; Diabetes Mellitus
Keywords: Heart Failure, Diabetes Mellitus, Mitochondrial Respiration
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Myocardial biopsies blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Control
- Insulin Resistant: Insulin Resistant
- Type 2 Diabetes: Type 2 Diabetes

SUMMARY:
Assessment of cardiac energy metabolism in patients with impaired glucose tolerance

DETAILED DESCRIPTION:
Insulin resistance, hepatocellular lipids (HCL) and plasma concentrations of free fatty acids (FFA) are predictors of heart failure, the leading cause of mortality in patients suffering from type 2 diabetes mellitus (T2DM). Epidemiological data suggest that diabetic cardiomyopathy (DC) presents as ventricular dysfunction in patients with T2DM independent of coronary artery disease. The underlying cellular mechanisms are poorly understood. Reduced mitochondrial activity and insulin resistance of skeletal muscle relates to liver steatosis, possibly due to higher substrate flux to the liver. High oxidation rates in the liver result in oxidative stress, damage of mitochondria and apoptosis. The investigators hypothesize that (i) HCL and impaired liver energy metabolism correlate with ventricular dysfunction, (ii) impaired glucose uptake and mitochondrial capacity in skeletal muscle relates to enhanced oxidative capacity, oxidative stress and lipid deposition in heart tissue (iii) reduced myocardial oxidative capacity limits recovery of myocardial function in patients with acute heart failure.

The investigators aim to assess (i) liver energy metabolism and heart function, (ii) respiration and lipid metabolites in skeletal muscle and heart tissue in humans with advanced heart failure and (iii) the prognostic impact of these factors in humans with acute heart failure.

This study will improve the understanding of mechanisms underlying the development of DC and the identification of patients at risk for poor outcome in heart failure.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20 and ≤85 years
* myocardial biopsy for medical reason

Exclusion Criteria:

* acute infection
* autoimmune disease
* pregnancy
* cancer

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing myocardial biopsy, left ventricular assist device implantation or heart transplantation for medical reasons
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
mitochondrial oxygen flux | Up to 36 months
  measured using high resolution respirometry. Unit: pmol/(s*mg)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Szendroedi, Prof., MD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zweck E, Scheiber D, Jelenik T, Bonner F, Horn P, Pesta D, Schultheiss HP, Boeken U, Akhyari P, Lichtenberg A, Kelm M, Roden M, Westenfeld R, Szendroedi J. Exposure to Type 2 Diabetes Provokes Mitochondrial Impairment in Apparently Healthy Human Hearts. Diabetes Care. 2021 May;44(5):e82-e84. doi: 10.2337/dc20-2255. No abstract available. PMID 33972315
- [Derived] Jelenik T, Flogel U, Alvarez-Hernandez E, Scheiber D, Zweck E, Ding Z, Rothe M, Mastrototaro L, Kohlhaas V, Kotzka J, Knebel B, Muller-Wieland D, Moellendorf S, Godecke A, Kelm M, Westenfeld R, Roden M, Szendroedi J. Insulin Resistance and Vulnerability to Cardiac Ischemia. Diabetes. 2018 Dec;67(12):2695-2702. doi: 10.2337/db18-0449. Epub 2018 Sep 26. PMID 30257974